CLINICAL TRIAL: NCT02348476
Title: A Study of Simbrinza™ Therapy in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-SIM-14-024
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Simbrinza™: Patients treated with Simbrinza™ (brinzolamide 1%/brimonidine 0.2%) as standard of care in clinical practice. No study drug is administered in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No study drug is administered in this study.

SUMMARY:
This study is a retrospective chart review to assess the tolerability and efficacy of treatment with Simbrinza™ used for patients with Open-Angle Glaucoma or Ocular Hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Participants treated with Simbrinza™ for Intra-Ocular Pressure (IOP) lowering in at least one eye
* Participants who had at least one-follow-up visit with tolerablity and efficacy data after Simbrinza™ treatment initiation.

Exclusion criteria:

* Active ocular disease other than glaucoma or ocular hypertension
* History of any intraocular surgery or glaucoma laser surgery within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Open-Angle Glaucoma or Ocular Hypertension treated in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The time to first glaucoma therapy escalation occurrence or discontinuation of Simbrinza® | 2 Years

SECONDARY OUTCOMES:
The time to first glaucoma therapy escalation occurrence | 2 Years
The time(s) to additional glaucoma therapy escalation occurrence(s) | 2 Years
Specific AEs and SAEs occurring with a frequency of ≥5% | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Wheaton, Illinois, United States